CLINICAL TRIAL: NCT04906070
Title: Study of the Safety and Efficacy of Radiation Therapy (HB-001) by Alpha-particle Sources for Recurrent Malignant Solid Tumors in Japan
Brief Title: Radiation Therapy (HB-001) by Alpha-particle Sources for Recurrent Malignant Solid Tumors in Japan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hekabio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HB-AT-001
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer; Head and Neck Cancer
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HB-001 DaRT Seeds (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seeds
  Interventions: Device: HB-001

INTERVENTIONS:
Device: HB-001 — An intratumoral insertion of a seed(s), loaded with Radium-224, securely fixed in the seeds. The seeds release by recoil into the tumor short-lived alpha-emitting atoms.
  Other Names: DaRT(Diffusing Alpha Radiation Emitters Therapy)

SUMMARY:
An intratumoral alpha particle based approach for cancer treatment using diffusion alpha-emitting radiation therapy (DaRT)

DETAILED DESCRIPTION:
This will be a prospective, open label, single arm, controlled study, assessing the safety and efficacy of diffusing alpha emitters radiation therapy (DaRT) delivered through radioactive seeds inserted into the tumor. This approach combines the advantages of local intratumoral irradiation of the tumor, as used in conventional brachytherapy, with the power of the alpha radiation emitting atoms, that will be introduced in quantities considerably lower than radiation therapy already used in patients. Superficial lesions with histopathological confirmation of malignancy will be treated using DaRT seeds. Reduction in tumor size 70 days after DaRT insertion will be assessed. Safety will be assessed by the incidence, severity and frequency of all Adverse Events (AE).

ELIGIBILITY:
Inclusion Criteria:

1. Head and neck cancer or breast cancer patients with histopathological proven malignancies who have a history of radiation therapy and who have been diagnosed with refractory malignancies with or without medical treatment.
2. Tumor size is 5 cm or less in the longest diameter
3. Age 18 years or older
4. Eastern Cooperative Oncology Group performance status is 2 or less
5. Life expectancy: 6 months or longer
6. Vital signs (systolic and diastolic blood pressure, pulse rate, body temperature, and respiratory rate) are stable
7. Platelet count >= 100,000/mm3 and prothrombin time Prothrombin Time-International Normalized Ratio <= 1.8
8. Women of childbearing potential have to be confirmed not pregnant by a pregnancy test and have to agree to prevent conception throughout the study.
9. Having received explanation about the study, consented to participate in the study and signed the informed consent form.
10. Measurable disease according to RECIST v1.1

Exclusion Criteria:

1. The size of the tumor more than 5 cm in the maximum diameter.
2. ECOG performance status is 3 or higher
3. Continuously receiving medication that may have a significant impact on the evaluation of safety or efficacy, such as immunosuppressants and/or corticosteroids.
4. History of serious allergy to the medicine for the treatments like anesthesia.
5. There are tumors to be preferentially treated such as metastatic lesion other than the target tumor
6. Having received chemotherapeutic drugs (except hormonal agents), immunotherapeutic agents, and molecular targeting agents in the past 30 days, which may affect the assessment of the safety or efficacy of the HB-001 brachytherapy.
7. Having received immune checkpoint inhibitor in the past 2 months, which may affect the assessment of the safety or efficacy of the HB-001 brachytherapy.
8. Having participated in different clinical studies in the past 30 days, which may affect the assessment of the safety or efficacy of HB-001 brachytherapy
9. Pregnant women or breast-feeding mothers
10. Those who do not wish to sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-05-25 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Tumor response to HB-001 | 9 - 11 weeks after HB-001 seed insertion
  Assessment of tumors response using the Response Evaluation Criteria in Solid Tumors (RECIST) (Version 1.1)

SECONDARY OUTCOMES:
Adverse Events | 12 weeks after HB-001 insertion
  The incidence, frequency, severity and causality of adverse events related to the HB-001

CONTACTS AND LOCATIONS:
Overall Officials: Toshiro Mabuchi, Study Director — Hekabio
Locations (4):
- Japan (4):
  - Tohoku University Hospital, Miyagi
  - Kansai Medical University Hospital, Osaka
  - National Cancer Center Hospital, Tokyo
  - Tokyo Medical And Dental University Medical Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No